CLINICAL TRIAL: NCT02560831
Title: Assessment of the Effects of Therapeutic Exercises Associated With Pompage Technique on Pain, Muscle Strength and Postural Balance in Older Women With Knee Osteoarthritis: a Randomized Clinical Trial
Brief Title: Effects of Therapeutic Exercises in Elderly Women With Knee Osteoarthritis
Acronym: TherExercOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Marcia Alessandra Carneiro Pedrosa de Castro, Profa. Dra., Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 02993812.3.0000.5208
Record Dates: First submitted 2015-09-22; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Therapeutic exercises; Pain; Muscle strength; Postural balance
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Therapeutic exercise and Pompage (Experimental): strengthening exercises, balance training and knee's pompage
  Interventions: Behavioral: Therapeutic exercise and Pompage
- Control (Active Comparator): Educational lectures.
  Interventions: Behavioral: Educational lectures

INTERVENTIONS:
Behavioral: Therapeutic exercise and Pompage — Strengthening exercises for flexors and knee extensors, balance training, knee's pompage twice per week for 12 weeks.
  Arms: Therapeutic exercise and Pompage
Behavioral: Educational lectures — Educational lectures in four meetings for 12 weeks (Control Group)
  Arms: Control

SUMMARY:
Knee Osteoarthritis is a degenerative disease associated with muscle weakness, arthralgia, rigidity and postural instability. Therapeutic exercise can reduce pain and improve muscle strength and postural balance, however benefits from association with pompage is not known. This study aims to evaluate the effects of therapeutic exercise on pain, muscle strength and postural balance in elderly women with knee osteoarthritis. Methodology: Almost randomized controlled trial, in which were included elderly between 60 and 80 years diagnosed with knee osteoarthritis, randomized into two groups with 11 participants each. Intervention group held strengthening exercises for flexors and knee extensors, balance training, and manual knee pompage for 12 weeks. Control Group received educational lectures. Arthralgia was estimated by pain subscale of the questionnaire Western Ontario McMaster Universities Osteoarthritis Index and (WOMAC); muscle strength was assessed by the isokinetic dynamometer HUMAC® NORM Testing & Rehabilitation System and the postural balance by the Biodex Balance SD postural stability protocol (Biodex Medical Systems, Inc. New York, USA). The Student t test was used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged between 60 and 80 years
* Diagnosed with knee's osteoarthritis according to clinical and radiographic criteria of the American College of Rheumatology.

Exclusion Criteria:

* Cardiovascular and/or unstable respiratory diseases
* Knee or hip arthroplasty; in the last 6 months: surgery on lower limbs, intraarticular corticosteroid injection in the knee, physical therapy
* Associated diseases that contribute to the balance disorders (for example ankylosing spondylitis, rheumatoid arthritis, diabetes mellitus, neurological diseases, Parkinson's disease, cerebral palsy and vestibular).

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The concentric muscular peak torque of the knee extensors | 3 months
  By isokinetic dynamometer HUMAC® NORM Testing & Rehabilitation System. It was rated the peak concentric muscle torque of knee extensors of both lower limbs at the speed of 120º/s. Patients were instructed to perform the knee extension at maximum amplitude pain-free permitted, then the maximum pain-free range in flexion. Movements of extension and flexion were performed five times for the participants to familiarize themselves with the procedure before the test. Then, five replicates were performed, and the highest amount recorded as peak muscle torque. All data were corrected by gravity. The values recorded in Newton-meters (Nm) were adjusted for body weight (kg) and presented as a percentage. For better analysis of peak concentric muscle torque of the knee extensors, the more symptomatic knee was assessed using the Visual Analogue Scale (VAS).
Postural stability | 3 months
  We used the Postural Stability Protocol, bipedal evaluation, eyes open eight resistance level and three repetitions of 20s with 10s rest. To mark the position of the feet, was adopted as the reference line of the heel and toe of the average tendon. The patient is positioned in front of a monitor containing a target and a cursor and Postural Stability protocol information. The therapist effected verbal command for the patient to keep a point at the center of the target, in which a lowest score (least deviation from the center) was desirable. The hand support or withdrawal of the platform legs was not allowed. Before the test, a simulation of the procedure was performed.

SECONDARY OUTCOMES:
Level of knee's pain | 3 months
  Was estimated by pain subscale of the questionnaire Western Ontario McMaster Universities Osteoarthritis Index and (WOMAC). This questionnaire consists of three domains: pain (5 questions), stiffness (2 questions) and functionality (17 questions), whose questions are answered by the volunteer about their perception in the last 72 hours. Higher scores indicate worse pain frame, rigidity or functionality. In our study, we used the score of the WOMAC pain questionnaire section. The items were evaluated levels: none, low, moderate, severe and very intense. For data analysis, the levels were calculated using a Likert 5-point scale: 0, 25, 50, 75 and 100.